CLINICAL TRIAL: NCT06736964
Title: Clinical Evaluation of Different Bioactive Restorative Materials for Cervical Carious in High Caries Risk Patients :A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Different Bioactive Restorative Materials for Cervical Carious in High Caries Risk Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yehia Hafez Yehia, Lecturer of Conservative Dentistry Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahmed abdul monsif
Record Dates: First submitted 2024-11-25; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Class V Dental Caries; High Caries Risk Patients
Keywords: bioactive restorative material; dual cure bulk fill bio-active restoration; Pre-reacted glass ionomer (PRG) Giomer

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double ( participant, Outcome Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Predicta (Experimental): based on dual cure bulk fill bioactive restoration
  Interventions: Device: Giomer
- Activa presto (Experimental): based on Bio-glass reinforced glass Ionomer
  Interventions: Device: Giomer
- Giomer (Active Comparator): based on Pre-reacted glass ionomer (PRG)
  Interventions: Device: Giomer

INTERVENTIONS:
Device: Giomer — based on Pre-reacted glass ionomer (PRG)

SUMMARY:
The aim of the study is to clinically evaluate three different bioactive restorative material in cervical carious lesion in high caries risk patients.

Reducing the incidence of recurrent caries is the primary outcome

DETAILED DESCRIPTION:
Bioactive restorative materials are relatively new concept in dentistry combines between esthetics, strength and resilience of composites with bioactive properties, the development of therapeutic bio-interactive materials results in tissue re-mineralization, reduces the susceptibility to tooth mineral loss, and recovers its mechanical properties .

Patients, with high caries, have many risk factors like inadequate biofilm control, salivary flow deficiency, and altered host defense. Conventional restorative materials expose the tooth structure to stress concentration. Moreover, preserving the tooth restoration interface intact is great challenge to avoid recurrent caries, which may also result in restoration failures .

This prospective study will be investigating and comparing the eighteen month clinical performance of a different bioactive restorative materials and a conventional Pre-reacted glass ionomer restorative material in class V cavity preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patient age range from 25-45 year.
* High risk caries.
* Patients required at least a couple of Class V restorations.
* The depth of lesion should be(1.5- 2 mm) .
* The patient should have good general health

Exclusion Criteria:

* Poor oral hygiene.
* Sever or chronic periodontal disease or Bruxism.
* Severe tooth sensitivity.
* Non-vital or fracture or cracked teeth.
* Defective restorations, orthodontic treatment or bleaching procedures during the last 6 months.
* pregnancy, and/or lactation, and allergy to the main components of the products to be used in the study

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
clinical performance (Post operative hyper sensitivity) | 12 months
  method of measurement is Modified United State Public Health Service Criteria (Modified USPHS) using Binary (yes/ no) yes outcome mean recurrent caries present, no mean no recurrent caries present .

SECONDARY OUTCOMES:
clinical performance (Fracture and retention, marginal integrity, marginal discoloration, anatomic form, surface texture, postoperative sensitivity) | 18 months
  method of measurement is Modified United State Public Health Service Criteria (Modified USPHS) using (Alpha ,Bravo, Charlie) as unite of measurement by scoring %.
  Alpha is best outcome and Charlie worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Nasr, professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
all collected IPD will be shared with supervisor: dr.Ashraf Nasr , Dr. yahia Hafez

DOCUMENTS (3):
  • Study Protocol (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT06736964/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT06736964/SAP_001.pdf
  • Informed Consent Form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT06736964/ICF_002.pdf